CLINICAL TRIAL: NCT06239831
Title: Postoperative Respiratory and Activity Monitoring
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22-2268
Record Dates: First submitted 2023-09-28; First posted 2024-02-02 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hypoventilation; Hypoxemia; Postoperative Pulmonary Complications
Keywords: hypoventilation; postoperative activity; abdominal surgery; mobilization; predicted minute ventilation (MVPred); accelerometer; chest monitor; postoperative pulmonary complications; surgical outcomes
MeSH Terms: conditions — Hypoventilation; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Postoperative monitoring: ActivPAL accelerometer will be placed on the chest and thigh, an ExSpiron monitor placed on the chest, and the patient will be observed for three days, until fully ambulatory (able to walk 30 meters without assistance with or without a walker), or until discharge; whichever comes earlier.
  Interventions: Device: ExSpiron and ActivPAL Monitors

INTERVENTIONS:
Device: ExSpiron and ActivPAL Monitors — ExSpiron chest monitor will be placed on the chest ActivPAL accelerometer will be placed on the chest and thigh

SUMMARY:
This study plans to learn more about specific breathing and activity recommendations for patients after surgery. Participants will be monitored after abdominal surgery to identify what activities help them breathe better and reduce complications after surgery.

DETAILED DESCRIPTION:
Investigators will study adults undergoing elective abdominal surgery with at least moderate risk for postoperative pulmonary complications.

Participants will be monitored on their chest and thigh with devices that record their breathing pattern (breath volume and frequency) and body position and movements. These monitors will be placed on their skin in the Post-Anesthesia Care Unit (PACU) and will stay on for three days, or until the patient is able to ambulate freely or until their hospital discharge, whichever comes earlier. Investigators will analyze the association between the frequency, duration and intensity of various activities (e.g., sitting, walking) and breathing and other clinical complications, in combination with medications received and other hospital course events.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 or older
* Must be undergoing abdominal surgery
* Must be high-risk for PPCs (ARISCAT score equal to or greater than 26)

Exclusion Criteria:

* Anyone under 18
* Anyone not undergoing abdominal surgery
* Anyone that is not high-risk for PPCs (ARISCAT score less than 26)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 undergoing abdominal surgery at the University of Colorado Health Hospital (UCHealth) that it high-risk for postoperative pulmonary complications (PPCs).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Hypoventilation | First 3 postoperative days
  Minutes per hour of hypoventilation which is defined as <40% of a predicted minute ventilation volume

SECONDARY OUTCOMES:
Variability of MV | Through postoperative day 3
  Variability of minute ventilation (MV)
Variability of VT | Through postoperative day 3
  Variability of tidal volume (VT)
Variability of RR | Through postoperative day 3
  Variability of respiratory rate (RR)
Events of Low MV | Through postoperative day 3
  Total number of events of low minute ventilation (MV)
Events of Low VT | Through postoperative day 3
  Total number of events of low tidal volume (VT)
Events of Low RR | Through postoperative day 3
  Total number of events of low respiratory rate (RR)
Percentage of time free of low or high MV | Through postoperative day 3
  The percentage of hours per day free of any low or high minute ventilation (MV)
Percentage of time free of low or high VT | Through postoperative day 3
  The percentage of hours per day free of any low or high tidal volume (VT)
Percentage of time free of low or high RR | Through postoperative day 3
  The percentage of hours per day free of any low or high resting rate (RR).
Duration of low MV | Through postoperative day 3
  Duration of low minute ventilation (MV)
Duration of low VT | Through postoperative day 3
  Duration of low tidal volume (VT)
Duration of low RR | Through postoperative day 3
  Duration of low respiratory rate (RR)
Duration of high MV | Through postoperative day 3
  Duration of low or high minute ventilation (MV)
Duration of high TV | Through postoperative day 3
  Duration of high tidal volume (VT)
Duration of high RR | Through postoperative day 3
  Duration of high respiratory rate (RR)
Postoperative Pulmonary Complication (PPC) Incidence | Through postoperative day 7
  Incidence of Postoperative Pulmonary Complications, or PPCs
Postoperative Pulmonary Complication (PPC) Severity | Through postoperative day 7
  Postoperative Pulmonary Complications, or PPCs, will be observed in their severity. PPC severity is defined as the most serious from Grade 0 (none) to Grade 4 (severe)
Time After Surgery to Sitting | Through postoperative day 3
  Time it takes for the patient to sit in a chair after surgery
Time After Surgery to Ambulating | Through postoperative day 3
  Time it takes for the patient to ambulate with and without help
Total Minutes Walking | Through postoperative day 3
  Patient's total minutes of walking
Total Walking Distance | Through postoperative day 3
  Patient's total walking distance (in meters)
Frequency of Ambulation | Through postoperative day 3
  How many times the patient gets up to ambulate
Time Spent in Bed | Through postoperative day 3
  After the surgery, the patient's minutes spent in bed
Time Spent in Sitting | Through postoperative day 3
  After the surgery, the patient's minutes spent sitting
Time Spent Standing | Through postoperative day 3
  After the surgery, the patient's minutes spent standing
Time Spent Walking | Through postoperative day 3
  After the surgery, the patient's minutes spent walking
Average Speed of Ambulation | Through postoperative day 3
  After the surgery, the patient's average speed of ambulating
First Postoperative Day Achieving Independent Ambulation | Through postoperative day 3
  After the surgery, the patient's first day of ambulating by his or herself for 30 meters
Metabolic Equivalent of Task (MET) Score of Physical Activity | Through postoperative day 3
  After the surgery, the patient's intensity of physical activity measured in METs
Other complications | Through postoperative day 7
  Incidence of any non-respiratory complications
Adverse events | Through postoperative day 7
  Incidence of any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fernandez-Bustamante, MD, PhD, Principal Investigator — University of Colorado Anschutz Medical Campus, University of Colorado Health Hospital
Locations (1):
- UC Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Bustamante A, Parker RA, Sprung J, Eikermann M, Gama de Abreu M, Ferrando C, Thompson BT, Vidal Melo MF. An anesthesia-centered bundle to reduce postoperative pulmonary complications: The PRIME-AIR study protocol. PLoS One. 2023 Apr 6;18(4):e0283748. doi: 10.1371/journal.pone.0283748. eCollection 2023. PMID 37023031
- [Background] Lawrence VA, Hilsenbeck SG, Mulrow CD, Dhanda R, Sapp J, Page CP. Incidence and hospital stay for cardiac and pulmonary complications after abdominal surgery. J Gen Intern Med. 1995 Dec;10(12):671-8. doi: 10.1007/BF02602761. PMID 8770719
- [Background] Fernandez-Perez ER, Sprung J, Afessa B, Warner DO, Vachon CM, Schroeder DR, Brown DR, Hubmayr RD, Gajic O. Intraoperative ventilator settings and acute lung injury after elective surgery: a nested case control study. Thorax. 2009 Feb;64(2):121-7. doi: 10.1136/thx.2008.102228. Epub 2008 Nov 6. PMID 18988659
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Shander A, Fleisher LA, Barie PS, Bigatello LM, Sladen RN, Watson CB. Clinical and economic burden of postoperative pulmonary complications: patient safety summit on definition, risk-reducing interventions, and preventive strategies. Crit Care Med. 2011 Sep;39(9):2163-72. doi: 10.1097/CCM.0b013e31821f0522. PMID 21572323
- [Background] Nijbroek SG, Schultz MJ, Hemmes SNT. Prediction of postoperative pulmonary complications. Curr Opin Anaesthesiol. 2019 Jun;32(3):443-451. doi: 10.1097/ACO.0000000000000730. PMID 30893115
- [Background] Kor DJ, Lingineni RK, Gajic O, Park PK, Blum JM, Hou PC, Hoth JJ, Anderson HL 3rd, Bajwa EK, Bartz RR, Adesanya A, Festic E, Gong MN, Carter RE, Talmor DS. Predicting risk of postoperative lung injury in high-risk surgical patients: a multicenter cohort study. Anesthesiology. 2014 May;120(5):1168-81. doi: 10.1097/ALN.0000000000000216. PMID 24755786
- [Background] Sabate S, Mazo V, Canet J. Predicting postoperative pulmonary complications: implications for outcomes and costs. Curr Opin Anaesthesiol. 2014 Apr;27(2):201-9. doi: 10.1097/ACO.0000000000000045. PMID 24419159
- [Background] Brueckmann B, Villa-Uribe JL, Bateman BT, Grosse-Sundrup M, Hess DR, Schlett CL, Eikermann M. Development and validation of a score for prediction of postoperative respiratory complications. Anesthesiology. 2013 Jun;118(6):1276-85. doi: 10.1097/ALN.0b013e318293065c. PMID 23571640
- [Background] LAS VEGAS investigators. Epidemiology, practice of ventilation and outcome for patients at increased risk of postoperative pulmonary complications: LAS VEGAS - an observational study in 29 countries. Eur J Anaesthesiol. 2017 Aug;34(8):492-507. doi: 10.1097/EJA.0000000000000646. PMID 28633157
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Milot J, Perron J, Lacasse Y, Letourneau L, Cartier PC, Maltais F. Incidence and predictors of ARDS after cardiac surgery. Chest. 2001 Mar;119(3):884-8. doi: 10.1378/chest.119.3.884. PMID 11243972
- [Background] Blum JM, Stentz MJ, Dechert R, Jewell E, Engoren M, Rosenberg AL, Park PK. Preoperative and intraoperative predictors of postoperative acute respiratory distress syndrome in a general surgical population. Anesthesiology. 2013 Jan;118(1):19-29. doi: 10.1097/ALN.0b013e3182794975. PMID 23221870
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Background] Bartels K, Kaizer A, Jameson L, Bullard K, Dingmann C, Fernandez-Bustamante A. Hypoxemia Within the First 3 Postoperative Days Is Associated With Increased 1-Year Postoperative Mortality After Adjusting for Perioperative Opioids and Other Confounders. Anesth Analg. 2020 Aug;131(2):555-563. doi: 10.1213/ANE.0000000000004553. PMID 31971921
- [Background] Bojesen RD, Fitzgerald P, Munk-Madsen P, Eriksen JR, Kehlet H, Gogenur I. Hypoxaemia during recovery after surgery for colorectal cancer: a prospective observational study. Anaesthesia. 2019 Aug;74(8):1009-1017. doi: 10.1111/anae.14691. Epub 2019 May 17. PMID 31099028
- [Background] Belcher AW, Khanna AK, Leung S, Naylor AJ, Hutcherson MT, Nguyen BM, Makarova N, Sessler DI, Devereaux PJ, Saager L. Long-Acting Patient-Controlled Opioids Are Not Associated With More Postoperative Hypoxemia Than Short-Acting Patient-Controlled Opioids After Noncardiac Surgery: A Cohort Analysis. Anesth Analg. 2016 Dec;123(6):1471-1479. doi: 10.1213/ANE.0000000000001534. PMID 27607476
- [Background] Zeng C, Lagier D, Lee JW, Vidal Melo MF. Perioperative Pulmonary Atelectasis: Part I. Biology and Mechanisms. Anesthesiology. 2022 Jan 1;136(1):181-205. doi: 10.1097/ALN.0000000000003943. PMID 34499087
- [Background] Hedenstierna G, Edmark L. Mechanisms of atelectasis in the perioperative period. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):157-69. doi: 10.1016/j.bpa.2009.12.002. PMID 20608554
- [Background] Brooks-Brunn JA. Postoperative atelectasis and pneumonia: risk factors. Am J Crit Care. 1995 Sep;4(5):340-9; quiz 350-1. PMID 7489036
- [Background] Hewlett AM, Branthwaite MA. Postoperative pulmonary function. Br J Anaesth. 1975 Feb;47(2):102-7. doi: 10.1093/bja/47.2.102. No abstract available. PMID 1096910
- [Background] Zwillich C, Kryger M, Weil J. Hypoventilation: consequences and management. Adv Intern Med. 1978;23:287-306. No abstract available. PMID 343542
- [Background] Craig DB, Wahba WM, Don HF, Couture JG, Becklake MR. "Closing volume" and its relationship to gas exchange in seated and supine positions. J Appl Physiol. 1971 Nov;31(5):717-21. doi: 10.1152/jappl.1971.31.5.717. No abstract available. PMID 5117187
- [Background] Noba L, Rodgers S, Chandler C, Balfour A, Hariharan D, Yip VS. Enhanced Recovery After Surgery (ERAS) Reduces Hospital Costs and Improve Clinical Outcomes in Liver Surgery: a Systematic Review and Meta-Analysis. J Gastrointest Surg. 2020 Apr;24(4):918-932. doi: 10.1007/s11605-019-04499-0. Epub 2020 Jan 3. PMID 31900738
- [Background] Ripolles-Melchor J, Ramirez-Rodriguez JM, Casans-Frances R, Aldecoa C, Abad-Motos A, Logrono-Egea M, Garcia-Erce JA, Camps-Cervantes A, Ferrando-Ortola C, Suarez de la Rica A, Cuellar-Martinez A, Marmana-Mezquita S, Abad-Gurumeta A, Calvo-Vecino JM; POWER Study Investigators Group for the Spanish Perioperative Audit and Research Network (REDGERM). Association Between Use of Enhanced Recovery After Surgery Protocol and Postoperative Complications in Colorectal Surgery: The Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol (POWER) Study. JAMA Surg. 2019 Aug 1;154(8):725-736. doi: 10.1001/jamasurg.2019.0995. PMID 31066889
- [Background] Lillemoe HA, Aloia TA. Enhanced Recovery After Surgery: Hepatobiliary. Surg Clin North Am. 2018 Dec;98(6):1251-1264. doi: 10.1016/j.suc.2018.07.011. Epub 2018 Aug 24. PMID 30390857
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Castelino T, Fiore JF Jr, Niculiseanu P, Landry T, Augustin B, Feldman LS. The effect of early mobilization protocols on postoperative outcomes following abdominal and thoracic surgery: A systematic review. Surgery. 2016 Apr;159(4):991-1003. doi: 10.1016/j.surg.2015.11.029. Epub 2016 Jan 21. PMID 26804821
- [Background] Lumb AB, Nunn JF. Respiratory function and ribcage contribution to ventilation in body positions commonly used during anesthesia. Anesth Analg. 1991 Oct;73(4):422-6. doi: 10.1213/00000539-199110000-00010. PMID 1897767
- [Background] Meyers JR, Lembeck L, O'Kane H, Baue AE. Changes in functional residual capacity of the lung after operation. Arch Surg. 1975 May;110(5):576-83. doi: 10.1001/archsurg.1975.01360110122020. PMID 1093513
- [Background] Ceylan B, Khorshid L, Gunes UY, Zaybak A. Evaluation of oxygen saturation values in different body positions in healthy individuals. J Clin Nurs. 2016 Apr;25(7-8):1095-100. doi: 10.1111/jocn.13189. Epub 2016 Feb 16. PMID 26879626
- [Background] Hardie JA, Morkve O, Ellingsen I. Effect of body position on arterial oxygen tension in the elderly. Respiration. 2002;69(2):123-8. doi: 10.1159/000056314. PMID 11961425
- [Background] van der Leeden M, Huijsmans R, Geleijn E, de Lange-de Klerk ES, Dekker J, Bonjer HJ, van der Peet DL. Early enforced mobilisation following surgery for gastrointestinal cancer: feasibility and outcomes. Physiotherapy. 2016 Mar;102(1):103-10. doi: 10.1016/j.physio.2015.03.3722. Epub 2015 May 7. PMID 26059985
- [Background] Haines KJ, Skinner EH, Berney S; Austin Health POST Study Investigators. Association of postoperative pulmonary complications with delayed mobilisation following major abdominal surgery: an observational cohort study. Physiotherapy. 2013 Jun;99(2):119-25. doi: 10.1016/j.physio.2012.05.013. Epub 2012 Sep 23. PMID 23219632
- [Background] Jonsson LR, Ingelsrud LH, Tengberg LT, Bandholm T, Foss NB, Kristensen MT. Physical performance following acute high-risk abdominal surgery: a prospective cohort study. Can J Surg. 2018 Feb;61(1):42-49. doi: 10.1503/cjs.012616. Epub 2017 Dec 1. PMID 29368676
- [Background] Cassidy MR, Rosenkranz P, McCabe K, Rosen JE, McAneny D. I COUGH: reducing postoperative pulmonary complications with a multidisciplinary patient care program. JAMA Surg. 2013 Aug;148(8):740-5. doi: 10.1001/jamasurg.2013.358. PMID 23740240
- [Background] Oliver CM, Warnakulasuriya S, McGuckin D, Singleton G, Martin P, Santos C, Bedford J, Wagstaff D, Sahni A, Gilhooly D, Wilson J, Edwards K, Baumber R, Vindrola-Padros C, Dorey J, Leeman I, Boyd-Carson H, Vohra R, Singh P, Bedford M, Vallance A, Aresu G, Tucker O, Swart M, Mythen MG; PQIP project delivery team; Moonesinghe SR; PQIP collaborative. Delivery of drinking, eating and mobilising (DrEaMing) and its association with length of hospital stay after major noncardiac surgery: observational cohort study. Br J Anaesth. 2022 Jul;129(1):114-126. doi: 10.1016/j.bja.2022.03.021. Epub 2022 May 12. PMID 35568508
- [Background] Grass F, Pache B, Martin D, Addor V, Hahnloser D, Demartines N, Hubner M. Feasibility of early postoperative mobilisation after colorectal surgery: A retrospective cohort study. Int J Surg. 2018 Aug;56:161-166. doi: 10.1016/j.ijsu.2018.06.024. Epub 2018 Jun 20. PMID 29935366
- [Background] Fiore JF Jr, Castelino T, Pecorelli N, Niculiseanu P, Balvardi S, Hershorn O, Liberman S, Charlebois P, Stein B, Carli F, Mayo NE, Feldman LS. Ensuring Early Mobilization Within an Enhanced Recovery Program for Colorectal Surgery: A Randomized Controlled Trial. Ann Surg. 2017 Aug;266(2):223-231. doi: 10.1097/SLA.0000000000002114. PMID 27997472
- [Background] Balvardi S, Pecorelli N, Castelino T, Niculiseanu P, Alhashemi M, Liberman AS, Charlebois P, Stein B, Carli F, Mayo NE, Feldman LS, Fiore JF Jr. Impact of Facilitation of Early Mobilization on Postoperative Pulmonary Outcomes After Colorectal Surgery: A Randomized Controlled Trial. Ann Surg. 2021 May 1;273(5):868-875. doi: 10.1097/SLA.0000000000003919. PMID 32324693
- [Background] Pottenger BC, Pronovost PJ, Kreif J, Klein L, Hobson D, Young D, Hoyer EH. Towards improving hospital workflows: An evaluation of resources to mobilize patients. J Nurs Manag. 2019 Jan;27(1):27-34. doi: 10.1111/jonm.12644. Epub 2018 Aug 16. PMID 30117210
- [Background] Schumann R, Kwater AP, Bonney I, Ladd D, Kim J, Gupta A, Gumbert SD, Pivalizza EG. Respiratory volume monitoring in an obese surgical population and the prediction of postoperative respiratory depression by the STOP-bang OSA risk score. J Clin Anesth. 2016 Nov;34:295-301. doi: 10.1016/j.jclinane.2016.04.029. Epub 2016 Jun 1. PMID 27687395
- [Background] Mehta JH, Cattano D, Brayanov JB, George EE. Assessment of perioperative minute ventilation in obese versus non-obese patients with a non-invasive respiratory volume monitor. BMC Anesthesiol. 2017 Apr 26;17(1):61. doi: 10.1186/s12871-017-0352-0. PMID 28446134
- [Background] Cella D, Choi SW, Condon DM, Schalet B, Hays RD, Rothrock NE, Yount S, Cook KF, Gershon RC, Amtmann D, DeWalt DA, Pilkonis PA, Stone AA, Weinfurt K, Reeve BB. PROMIS(R) Adult Health Profiles: Efficient Short-Form Measures of Seven Health Domains. Value Health. 2019 May;22(5):537-544. doi: 10.1016/j.jval.2019.02.004. PMID 31104731
- [Background] Atkinson DB, Sens BA, Bernier RS, Gomez-Morad AD, Imsirovic J, Nasr VG. The Evaluation of a Noninvasive Respiratory Volume Monitor in Mechanically Ventilated Neonates and Infants. Anesth Analg. 2022 Jan 1;134(1):141-148. doi: 10.1213/ANE.0000000000005562. PMID 33929346
- [Background] Gomez-Morad AD, Cravero JP, Harvey BC, Bernier R, Halpin E, Walsh B, Nasr VG. The Evaluation of a Noninvasive Respiratory Volume Monitor in Pediatric Patients Undergoing General Anesthesia. Anesth Analg. 2017 Dec;125(6):1913-1919. doi: 10.1213/ANE.0000000000002029. PMID 28759491
- [Background] Gonzalez Castro LN, Mehta JH, Brayanov JB, Mullen GJ. Quantification of respiratory depression during pre-operative administration of midazolam using a non-invasive respiratory volume monitor. PLoS One. 2017 Feb 24;12(2):e0172750. doi: 10.1371/journal.pone.0172750. eCollection 2017. PMID 28235069
- [Background] Ebert TJ, Middleton AH, Makhija N. Ventilation monitoring during moderate sedation in GI patients. J Clin Monit Comput. 2017 Feb;31(1):53-57. doi: 10.1007/s10877-015-9809-1. Epub 2015 Dec 1. PMID 26628270
- [Background] van den Bosch OFC, Alvarez-Jimenez R, Stam MMH, den Boer FC, Loer SA. Variations in respiratory rate do not reflect changes in tidal volume or minute ventilation after major abdominal surgery. J Clin Monit Comput. 2021 Aug;35(4):787-796. doi: 10.1007/s10877-020-00538-3. Epub 2020 Jun 1. PMID 32488678
- [Background] Williams GW 2nd, George CA, Harvey BC, Freeman JE. A Comparison of Measurements of Change in Respiratory Status in Spontaneously Breathing Volunteers by the ExSpiron Noninvasive Respiratory Volume Monitor Versus the Capnostream Capnometer. Anesth Analg. 2017 Jan;124(1):120-126. doi: 10.1213/ANE.0000000000001395. PMID 27384980
- [Background] O'Brien CM, Duda JL, Kitas GD, Veldhuijzen van Zanten JJCS, Metsios GS, Fenton SAM. Measurement of sedentary time and physical activity in rheumatoid arthritis: an ActiGraph and activPAL validation study. Rheumatol Int. 2020 Sep;40(9):1509-1518. doi: 10.1007/s00296-020-04608-2. Epub 2020 May 29. PMID 32472303
- [Background] Crowley P, Skotte J, Stamatakis E, Hamer M, Aadahl M, Stevens ML, Rangul V, Mork PJ, Holtermann A. Comparison of physical behavior estimates from three different thigh-worn accelerometers brands: a proof-of-concept for the Prospective Physical Activity, Sitting, and Sleep consortium (ProPASS). Int J Behav Nutr Phys Act. 2019 Aug 16;16(1):65. doi: 10.1186/s12966-019-0835-0. PMID 31419998
- [Background] Rosenberger ME, Buman MP, Haskell WL, McConnell MV, Carstensen LL. Twenty-four Hours of Sleep, Sedentary Behavior, and Physical Activity with Nine Wearable Devices. Med Sci Sports Exerc. 2016 Mar;48(3):457-65. doi: 10.1249/MSS.0000000000000778. PMID 26484953
- [Background] Lyden K, John D, Dall P, Granat MH. Differentiating Sitting and Lying Using a Thigh-Worn Accelerometer. Med Sci Sports Exerc. 2016 Apr;48(4):742-7. doi: 10.1249/MSS.0000000000000804. PMID 26516691
- [Background] Steeves JA, Bowles HR, McClain JJ, Dodd KW, Brychta RJ, Wang J, Chen KY. Ability of thigh-worn ActiGraph and activPAL monitors to classify posture and motion. Med Sci Sports Exerc. 2015 May;47(5):952-9. doi: 10.1249/MSS.0000000000000497. PMID 25202847
- [Background] Creasy SA, Crane TE, Garcia DO, Thomson CA, Kohler LN, Wertheim BC, Baker LD, Coday M, Hale L, Womack CR, Wright KP, Melanson EL. Higher amounts of sedentary time are associated with short sleep duration and poor sleep quality in postmenopausal women. Sleep. 2019 Jul 8;42(7):zsz093. doi: 10.1093/sleep/zsz093. PMID 30994175
- [Background] Ostendorf DM, Lyden K, Pan Z, Wyatt HR, Hill JO, Melanson EL, Catenacci VA. Objectively Measured Physical Activity and Sedentary Behavior in Successful Weight Loss Maintainers. Obesity (Silver Spring). 2018 Jan;26(1):53-60. doi: 10.1002/oby.22052. Epub 2017 Nov 1. PMID 29090513
- [Background] Carney MJ, Weissler JM, Fox JP, Tecce MG, Hsu JY, Fischer JP. Trends in open abdominal surgery in the United States-Observations from 9,950,759 discharges using the 2009-2013 National Inpatient Sample (NIS) datasets. Am J Surg. 2017 Aug;214(2):287-292. doi: 10.1016/j.amjsurg.2017.01.001. Epub 2017 Jan 12. PMID 28202162